CLINICAL TRIAL: NCT02071628
Title: Study for Validation of In-vitro Turbidometric Platelet Aggregation Assay Using Human Blood in Healthy Volunteers
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Kyun-Seop Bae, Asan Medical Center, Asan Medical Center
Other Study IDs: TGVT-1301
Record Dates: First submitted 2014-01-13; First posted 2014-02-26 (Estimated); Last update posted 2014-02-26 (Estimated); Status verified 2014-02

CONDITIONS: Validation of In-vitro Turbidometric Platelet Aggregation Assay

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This study is designed for validation of in-vitro platelet aggregation assay using human blood in healthy volunteers. 32ml blood, 2ml for complete blood count test and 30ml for platelet aggregation assay, was collected from ten subjects, respectively.

Preparation of Platelet Rich Plasma (PRP):

1. Collect human blood using 21g butterfly syringe and dilute 9:1 into 3.8% sodium citrate vacutainer vials.
2. Prepare platelet rich plasma (PRP) by centrifuging blood at 100 x g for 15 minutes at room temperature. Using a plastic transfer pipette, carefully transfer and combine PRP from multiple vacutainer tubes (if required) into a 15 mL conical tube.
3. PRP is removed re-centrifuge remaining blood in vacutainer tubes at 2000 x g for 15 minutes at room temp. to obtain platelet poor plasma (PPP). Transfer PPP to 15 mL conical tube.
4. Measure platelet count in combined PRP using Z1 Coulter Particle Counter or similar product. Adjust platelet count to a final concentration of 300,000 +- 10,000 platelets in PRP using PPP.

Aggregation Measurement:

Aggregation is measured using a model 490-X Chrono-Log Aggregometer or similar product. PPP is used as a reference to establish 100% optical transmission.

ELIGIBILITY:
Inclusion Criteria:

* 20-50years old
* must be able to consent voluntarily
* consent to keep the study terms of obedience

Exclusion Criteria:

* blood coagulation disorder or bleeding disorder
* blood donation within 60 days or blood transfusion within 30 days before screening
* smoker or who stopped smoking within 1month before screening
* administration of drugs such as anticoagulants or antiplatelets or alcohol within 14 days before screening
* eligibility failure under investigator's judgements

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy adult voulteers
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2013-12; Primary Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Maximal platelet aggregation(MPA) for the TRAP and 5-HT baseline aggregation response and the 5-HT amplification of TRAP-induced aggregation | Up to 6months
  Calculate each maximal platelet aggregation(MPA) for the TRAP and 5-HT baseline aggregation response and the 5-HT amplification of TRAP-induced aggregation, respectively. Compare the results with previous datas to evaluate the analysis machine and the assay methods.